CLINICAL TRIAL: NCT06308731
Title: A Crossover Study to Examine Exercise-Induced Rates of Fat Oxidation with and Without Ingestion of a Caffeine-Based Energy Drink
Brief Title: Exercise-Induced Rates of Fat Oxidation with and Without Ingestion of a Caffeine-Based Energy Drink
Acronym: EDX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lindenwood University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 23-26
Record Dates: First submitted 2023-12-08; First posted 2024-03-13 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Substrate Oxidation; Energy Expenditure; Reaction Time; Cognition; Exercise Performance
Keywords: energy drink; exercise performance

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo controlled, crossover design
Who Masked: Participant, Investigator
Masking Description: All energy drink supplements are provided in identical, unlabeled cans, using a randomization code.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Caffeine-Based Energy Drink (Experimental): 12 oz Caffeine-based energy drink providing 200 mg caffeine
  Interventions: Dietary Supplement: Caffeine-Based Energy Drink
- Placebo (Placebo Comparator): 12 oz placebo void of all active ingredients
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Caffeine-Based Energy Drink — Energy drink with 200 mg caffeine
  Arms: Caffeine-Based Energy Drink
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate acute changes in rates of fat oxidation during exercise with and without the ingestion of a caffeine-based energy drink.

DETAILED DESCRIPTION:
This study aims to investigate the impact of a caffeinated energy drink on cognitive function and exercise performance in healthy adults. The research will employ a randomized, double-blind, placebo-controlled, crossover design involving 15 participants. Initial screening includes health assessments and completion of a health history questionnaire, as well as a VO2peak assessment. Participants will replicate their diet before every study visit. Subsequent visits involve baseline assessments, ingestion of either a placebo or a caffeinated energy drink, followed by cognitive tests and a cycling exercise bout at moderate intensity, followed by a exercise performance cycling time trial. Measurements, including heart rate, perceived exertion, blood samples, and expired gases, will be collected during and after exercise. The study will have two identical testing visits, separated by at least a week, with participants consuming different beverages to assess their impact on cognitive function and exercise performance.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants between 18 - 50 years of age
* Signed informed consent
* Healthy defined as currently not being treated for an active cardiac, pulmonary, metabolic, immunological, neurological, respiratory, orthopedic, musculoskeletal, psychiatric, or reproductive disease or disorder. With the research team and principal investigator's discretion, some ongoing treatments will be permitted if a determination is made that the treatment will not increase the risk of study participation and the treatment will not confound with desired study outcomes
* Physically active which is defined as performing aerobic or resistance-based physical exercise between 2 and 5 times per week
* Moderate caffeine users (~300 mg/day)
* Body mass index values will range from >24.0 to < 31.9 kg/m2. The average body mass index for the entire study cohort will be less than 31.99 kg/m2. As such, an ongoing calculation of the recruited cohort's mean body mass index will be maintained and people will only be randomized into the study if the average cohort body mass index value does not exceed 31.99 kg/m2
* Willing and able to agree to the requirements and restrictions of this study, be willing to give voluntary consent, and carry out all study-related procedures

Exclusion Criteria:

* Body mass index > 31.9 kg/m2
* Positive medical history and/or is currently being treated for some form of heart or cardiovascular, neurological impairment, disease or condition, immune disorder or disease, thyroid disease, kidney disease, renal failure, regular dialysis, liver disease, or other diagnosed hepatic impairment
* Diagnosed with having Type I or Type II diabetes (determined as fasting blood glucose > 126 mg/dL)
* Diagnosed with major affective disorder or other psychiatric disorder that required hospitalization in the prior year
* History of cancer (except localized skin cancer without metastases or in situ cervical cancer within 5 years prior to screening visit).
* Participant has an abnormality or obstruction of the gastrointestinal tract precluding swallowing (e.g., dysphagia) and digestion (e.g., known intestinal malabsorption, celiac disease, inflammatory bowel disease, chronic pancreatitis, steatorrhea)
* Currently prescribed statin drugs (i.e., Lipitor, Livalo, Crestor, Zocor, etc.) or any hypertension medications (i.e., Beta-blockers, ACE Inhibitors, Alpha-blockers, Vasodilators, etc.) or any other medication at the discretion of the principal investigator
* Current smoker (>10 cigarettes per day)
* Participants who are lactating, pregnant, or planning to become pregnant
* History of alcohol or substance abuse in the 6 months prior to screening
* Receipt or use of an investigational product in another research study within 60 days of beginning the study protocol
* Any condition or abnormality that, in the opinion of the investigator, would compromise the safety of the participant or the quality of the study data
* Extensive travel (>1 month) that will disrupt the original outline of the study protocol

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2024-01-19 (Actual); Primary Completion 2024-09-16 (Actual); Study Completion 2024-09-16 (Actual)

PRIMARY OUTCOMES:
Impact of a caffeine-based energy drink ingestion on fat oxidation rates during exercise. | 150 minutes during exercise
  Fat oxidation rate (grams/min) during exercise

SECONDARY OUTCOMES:
Impact of a caffeine-based energy drink ingestion on energy expenditure rates during exercise. | 150 minutes during exercise
  Energy expenditure (kcals/min)
Impact of a caffeine-based energy drink ingestion on carbohydrate oxidation during exercise | 150 minutes during exercise
  Carbohydrate oxidation rates (grams/min)
Impact of a caffeine-based energy drink ingestion on plasma glycerol concentration | 150 minutes after intervention ingestion
  Plasma glycerol concentration
Impact of a caffeine-based energy drink ingestion on plasma free fatty acid concentration | 150 minutes after intervention ingestion
  Plasma free fatty acid concentration
Impact of a caffeine-based energy drink ingestion on ratings of perceived exertion | 150 minutes after intervention ingestion
  Rating of Perceived Exertion (RPE) scale
Impact of a caffeine-based energy drink ingestion on exercise performance | 150 minutes after intervention ingestion
  Cycling time trial
Impact of a caffeine-based energy drink ingestion on reaction time | 150 minutes after intervention ingestion
  Simple/ choice reaction time
Impact of a caffeine-based energy drink ingestion on trail making test performance | 150 minutes after intervention ingestion
  Trail making test
Impact of a caffeine-based energy drink ingestion on Cognition | 150 minutes after intervention ingestion
  Serial 7 Cognitive processing test

OTHER OUTCOMES:
Impact of a caffeine-based energy drink ingestion on adverse events | 3 weeks
  Self-reported adverse events
Impact of a caffeine-based energy drink ingestion on heart rate | 3 weeks
  Heart rate (bpm)
Impact of a caffeine-based energy drink ingestion on blood pressure | 3 weeks
  Blood Pressure (mmHg)

CONTACTS AND LOCATIONS:
Locations (1):
- Exercise and Performance Nutrition Laboratory, Saint Charles, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Investigators do not plan to make individual participant data available to other researchers